CLINICAL TRIAL: NCT06406972
Title: Brief Admission by Self-referral for Individuals With Self-harm: Effects on Compulsory Care
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Linkoeping University (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-02307-01
Record Dates: First submitted 2024-04-19; First posted 2024-05-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Self-injury; Suicide; Suicide, Attempted; Self-harm; Borderline Personality Disorder; Emergency Psychiatric; Hospitalizations Psychiatric
Keywords: Brief Admission by self-referral; self-harm; traits of borderline personality disorder; compulsory care
MeSH Terms: conditions — Self-Injurious Behavior; Suicide; Suicide, Attempted; Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Lund 2010-09-15-2015-09-14: Lund, before implementation of Brief Admission by self-referral
- Lund 2015-09-15-2020-09-14: Lund, after implementation of Brief Admission by self-referral in Lund, before implementation of Brief Admission by self-referral in Linköping
  Interventions: Other: Brief Admission by self-referral (BA)
- Lund 2020-09-15-2025-09-14: Lund, after implementation of Brief Admission by self-referral in Lund and in Linköping
  Interventions: Other: Brief Admission by self-referral (BA)
- Linköping 2010-09-15-2015-09-14: Linköping before implementation of Brief Admission by self-referral
- Linköping 2015-09-15-2020-09-14: Linköping after implementation of Brief Admission by self-referral in Lund, before implementation of Brief Admission by self-referral in Linköping
- Linköping 2020-09-15-2025-09-14: Linköping after implementation of Brief Admission by self-referral in Lund and in Linköping
  Interventions: Other: Brief Admission by self-referral (BA)
- Helsingborg 2014-02-15-2017-02-14: Helsingborg before implementation of Brief Admission by self-referral
- Helsingborg 2017-02-15-2020-02-14: Helsingborg after implementation of Brief Admission by self-referral in Helsingborg, before implementation of Brief Admission by self-referral in Norrköping
  Interventions: Other: Brief Admission by self-referral (BA)
- Helsingborg 2020-02-15-2023-02-14: Helsingborg after implementation of Brief Admission by self-referral in Helsingborg and in Norrköping
  Interventions: Other: Brief Admission by self-referral (BA)
- Norrköping 2014-02-15-2017-02-14: Norrköping before implementation of Brief Admission by self-referral
- Norrköping 2017-02-15-2020-02-14: Norrköping after implementation of Brief Admission by self-referral in Helsingborg, before implementation of Brief Admission by self-referral in Norrköping
- Norrköping 2020-02-15-2023-02-14: Norrköping after implementation of Brief Admission by self-referral in Helsingborg and in Norrköping
  Interventions: Other: Brief Admission by self-referral (BA)

INTERVENTIONS:
Other: Brief Admission by self-referral (BA) — Through means of an individualised contract access to self-referral to inpatient treatment limited to a maximum of three nights, three times per month.
  Other Names: Patient initiated Brief admission; Self-referral to inpatient treatment; Patient controlled hospital admission
  Groups: Helsingborg 2017-02-15-2020-02-14; Helsingborg 2020-02-15-2023-02-14; Linköping 2020-09-15-2025-09-14; Lund 2015-09-15-2020-09-14; Lund 2020-09-15-2025-09-14; Norrköping 2020-02-15-2023-02-14

SUMMARY:
Brief Admission by self-referral (BA) is a standardized treatment model, providing patient-controlled and person-centered care. It was developed to reduce self-harm and compulsory care by promoting autonomy. Randomized clinical trials have not yielded significant between group differences with respect to inpatient care, including compulsory care. The major difficulty in evaluating BA is preventing the control group from cross-contamination, as in the implementation process of BA, all physicians, all inpatient and outpatient staff as well as managers need to be informed and undergo basic education regarding the intervention. As BA addresses a prevalent and frustrating issue in psychiatric health care, there is considerable risk that the approach leaks to the control group, reducing the possibility to detect between-group differences. In the current study this will be addressed through a register-based approach, comparing similar clinics, implementing BA at different timepoints over time. Individuals with traits of borderline personality disorder will be included and comparisons will be made with respect to compulsory care, voluntary inpatient care and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Living in the uptake area of Lund, Linköping, Helsingborg or Norrköping
* Age 18-65 years at the time of inclusion
* Admitted to hospital either diagnosed with ICD-10 diagnosis BPD F60.3, or admitted at least twice with Intentional self-harm X60-83 in combination with one of more of the following diagnoses ADHD (F90.0-F90.X), Bipolar disorder type 2, (F31.8W, F318A-F, F31.0, F31.8-9, F31.8W) or Autism, Atypical autism, Aspergers syndrome (F84.0, F84.1, F84.5) or Mild intellectual disability (F70.0-F70.9).

Exclusion Criteria:

* not fulfilling inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with repeated self-harm and traits of Borderline personality disorder
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2010-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Days with compulsory admission | 2010-09-15 - 2025-09-14
  Days with compulsory admission (days/year)

SECONDARY OUTCOMES:
Days with voluntary psychiatric admission | 2010-09-15 - 2025-09-14
  Days with voluntary psychiatric admission (days/year)
Duration of free intervals between admissions | 2010-09-15 - 2025-09-14
  Duration of free intervals between admissions (days)
Mortality | 2010-09-15 - 2025-09-14
  All cause mortality as well as death by suicide specifically (X60-X84 and Y10-Y34 in ICD10)
Number of compulsory admissions | 2010-09-15 - 2025-09-14
  Number of compulsory admissions (admissions/year)
Number of voluntary psychiatric admissions (admissions/year) | 2010-09-15 - 2025-09-14
  Number of voluntary psychiatric admissions
Number of compulsory acts/year | 2010-09-15 - 2025-09-14
  Number of compulsory acts/year

OTHER OUTCOMES:
Gender distribution | 2010-09-15 - 2025-09-14
  Differences in distribution of diagnoses between men and women
Number of admissions with Brief admission by self-referral (BA) | 2010-09-15 - 2025-09-14
  Number of BA admissions (admissions/year)
Compulsory admission - median length | 2010-09-15 - 2025-09-14
  Compulsory admission - median length (days/admission)
Voluntary psychiatric admissions - median length | 2010-09-15 - 2025-09-14
  Voluntary psychiatric admissions - median length (days/admission)
Number of voluntary psychiatric admissions | 2010-09-15 - 2025-09-14
  Number of voluntary psychiatric admissions (admissions/year)

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Sofie, PhD, Principal Investigator — Lund University
Locations (4):
- Sweden (4):
  - Division of Psychiatry, Region Skåne, Lund, Skåne County
  - Region Östergötland, Linköping
  - Statistiska centralbyrån, Solna
  - Socialstyrelsen, Stockholm

REFERENCES:
- [Background] Warrender D. Borderline personality disorder and the ethics of risk management: The action/consequence model. Nurs Ethics. 2018 Nov;25(7):918-927. doi: 10.1177/0969733016679467. Epub 2017 Jan 19. PMID 28100114
- [Background] Coyle TN, Shaver JA, Linehan MM. On the potential for iatrogenic effects of psychiatric crisis services: The example of dialectical behavior therapy for adult women with borderline personality disorder. J Consult Clin Psychol. 2018 Feb;86(2):116-124. doi: 10.1037/ccp0000275. PMID 29369662
- [Background] Liljedahl SI, Helleman M, Daukantaite D, Westrin A, Westling S. A standardized crisis management model for self-harming and suicidal individuals with three or more diagnostic criteria of borderline personality disorder: The Brief Admission Skane randomized controlled trial protocol (BASRCT). BMC Psychiatry. 2017 Jun 15;17(1):220. doi: 10.1186/s12888-017-1371-6. PMID 28619050
- [Background] Strand M, von Hausswolff-Juhlin Y. Patient-controlled hospital admission in psychiatry: A systematic review. Nord J Psychiatry. 2015;69(8):574-86. doi: 10.3109/08039488.2015.1025835. Epub 2015 Apr 2. PMID 25832757
- [Background] Westling S, Daukantaite D, Liljedahl SI, Oh Y, Westrin A, Flyckt L, Helleman M. Effect of Brief Admission to Hospital by Self-referral for Individuals Who Self-harm and Are at Risk of Suicide: A Randomized Clinical Trial. JAMA Netw Open. 2019 Jun 5;2(6):e195463. doi: 10.1001/jamanetworkopen.2019.5463. PMID 31173128
- [Background] Lindkvist RM, Landgren K, Liljedahl SI, Daukantaite D, Helleman M, Westling S. Predictable, Collaborative and Safe: Healthcare Provider Experiences of Introducing Brief Admissions by Self-referral for Self-harming and Suicidal Persons with a History of Extensive Psychiatric Inpatient Care. Issues Ment Health Nurs. 2019 Jul;40(7):548-556. doi: 10.1080/01612840.2019.1585497. Epub 2019 May 17. PMID 31099707
- [Background] Sigrunarson V, Moljord IE, Steinsbekk A, Eriksen L, Morken G. A randomized controlled trial comparing self-referral to inpatient treatment and treatment as usual in patients with severe mental disorders. Nord J Psychiatry. 2017 Feb;71(2):120-125. doi: 10.1080/08039488.2016.1240231. Epub 2016 Oct 14. PMID 27739334
- [Background] Thomsen CT, Benros ME, Maltesen T, Hastrup LH, Andersen PK, Giacco D, Nordentoft M. Patient-controlled hospital admission for patients with severe mental disorders: a nationwide prospective multicentre study. Acta Psychiatr Scand. 2018 Apr;137(4):355-363. doi: 10.1111/acps.12868. Epub 2018 Mar 4. PMID 29504127

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT06406972/Prot_SAP_000.pdf